CLINICAL TRIAL: NCT01276314
Title: Evaluation of TNF-α Blockade Effect in Patients With Severe Cutaneous Adverse Drug Reactions (SCAR)
Brief Title: Evaluation of TNF-α Blockade Effect in Patients With Severe Cutaneous Adverse Drug Reactions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 97-1413A3
Record Dates: First submitted 2009-07-05; First posted 2011-01-13 (Estimated); Results first posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2014-12

CONDITIONS: Drug Hypersensitivity
Keywords: SCAR; anti-TNF-a
MeSH Terms: conditions — Drug Hypersensitivity; Cicatrix | interventions — Etanercept; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti- TNF-a treatment (Experimental): 1. Meet the conditions of inclusion and exclusion, seek the consent of the patient, and fill out the ICF
  2. Fill out the case report form
  3. Blood test and physiological assessment, and do TNF-alpha serum concentration and peripheral blood mononuclear spherical cDNA expression analysis
  4. Etanercept administration:
  The experimental group received the first dose of Etanercept (25 mg) i.v., followed by two doses per week and maintain 2 to 3 weeks
  Interventions: Drug: anti- TNF-a
- control group (Active Comparator): 1. Meet the conditions of inclusion and exclusion, seek the consent of the patient, and fill out the ICF
  2. Fill out the case report form
  3. Blood test and physiological assessment, and do TNF-alpha serum concentration and peripheral blood mononuclear spherical cDNA expression analysis
  4. Drug administration:
  The control group of drug delivery: systemic intravenous steroid therapy, the dose is equivalent to prednisolone 1-1.5 mg / kg / day, according to the treatment of 3-4 days gradually decreased dose.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: anti- TNF-a — 25mg BIW, SC
  Other Names: Etanercept
  Arms: anti- TNF-a treatment
Drug: Prednisolone — 1-1.5 mg / kg / day
  Other Names: steroid therapy
  Arms: control group

SUMMARY:
Severe skin adverse drug reactions can result in death. Toxic epidermal necrolysis (TEN) has the highest mortality (30-35%); Stevens-Johnson syndrome and transitional forms correspond to the same syndrome, but with less extensive skin detachment and a lower mortality (5-15%). Hypersensitivity syndrome, sometimes called Drug Reaction with Eosinophilia and Systemic Symptoms (DRESS), has a mortality rate evaluated at about 10%. The aims of this project are (1) to compare the effect of treatment between systemic steroid and anti-TNF-α. Including skin healing time, beginning of re-epithelialization time, internal organ recovery time, mortality rate, adverse events and (2) to investigate the molecular mechanism of severe cutaneous adverse reaction after anti-TNF-α treatment.

DETAILED DESCRIPTION:
Severe cutaneous adverse drug reactions, including Toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome(SJS), Drug Reaction with Eosinophilia and Systemic Symptoms (DRESS) is a life threatening disease. There is no gold standard in the therapy of SCAR. Treatment with high dose systemic corticosteroids is controversial. Although there have been recent reports of success with various therapies such as plasmapheresis and high-dose intravenous immunoglobulins, their efficacy is not yet proven. Assessment of these therapies is difficult because of their non-specific immunosuppressant or immunomodulating modes of action. Recent studies have shown evidence of the pathogenetic importance of tumour necrosis factor (TNF)-a, suggesting a new therapeutic approach in selective blockade of TNF-a using specific antibodies. We report successful treatment TEN using monoclonal IgG anti-TNF-antibodies. The aims of this project are (1) to compare the effect of treatment between systemic steroid and anti-TNF-α. Including skin healing time, beginning of re-epithelialization time, internal organ recovery time, mortality rate, adverse events and (2) to investigate the molecular mechanism of severe cutaneous adverse reaction after anti-TNF-α treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient with clinical and pathological diagnoses of severe cutaneous adverse drug reactions such as Stevens-Johnson Syndrome, Toxic Epidermal Necrolysis or Durg reaction with eosinophilia and systemic symptoms.
2. Male or female patient aged more than 4 years.
3. Inform consent obtained.

Exclusion Criteria:

1. Pregnant or breastfeeding female.
2. Allergic to any anti-TNF-α biological product.
3. Active or latent tuberculosis confirmed with Chest X-ray.
4. Severe active infection and septicemia.
5. Active Hepatitis B or C carrier.
6. Suspected HIV carrier with CD4 count less than 200.
7. Patient with poor compliance or with safety concerns judged by investigator.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2009-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Hung Chung, MD, Study Chair — Department of Dermatology, CGMH
Locations (1):
- Department of Dermatology, Chang Gung Memorial hospital, Taipei, Taiwan

REFERENCES:
- [Background] Paquet P, Paquet F, Al Saleh W, Reper P, Vanderkelen A, Pierard GE. Immunoregulatory effector cells in drug-induced toxic epidermal necrolysis. Am J Dermatopathol. 2000 Oct;22(5):413-7. doi: 10.1097/00000372-200010000-00005. PMID 11048976
- [Result] Schneck J, Fagot JP, Sekula P, Sassolas B, Roujeau JC, Mockenhaupt M. Effects of treatments on the mortality of Stevens-Johnson syndrome and toxic epidermal necrolysis: A retrospective study on patients included in the prospective EuroSCAR Study. J Am Acad Dermatol. 2008 Jan;58(1):33-40. doi: 10.1016/j.jaad.2007.08.039. Epub 2007 Oct 4. PMID 17919775
- [Result] Paradisi A, Abeni D, Bergamo F, Ricci F, Didona D, Didona B. Etanercept therapy for toxic epidermal necrolysis. J Am Acad Dermatol. 2014 Aug;71(2):278-83. doi: 10.1016/j.jaad.2014.04.044. Epub 2014 Jun 11. PMID 24928706
- [Derived] Wang CW, Yang LY, Chen CB, Ho HC, Hung SI, Yang CH, Chang CJ, Su SC, Hui RC, Chin SW, Huang LF, Lin YY, Chang WY, Fan WL, Yang CY, Ho JC, Chang YC, Lu CW, Chung WH; the Taiwan Severe Cutaneous Adverse Reaction (TSCAR) Consortium. Randomized, controlled trial of TNF-alpha antagonist in CTL-mediated severe cutaneous adverse reactions. J Clin Invest. 2018 Mar 1;128(3):985-996. doi: 10.1172/JCI93349. Epub 2018 Feb 5. PMID 29400697

RESULTS

PARTICIPANT FLOW:
Recruitment Details: SCAR patients were enrolled in the clinical trial from 2009 to 2015 at Chang Gung Memorial Hospital in Taiwan.
Pre-assignment Details: We totally recruited 140 participants, but only 135 SCAR participants (including 91 SJS/TEN patients and 44 DRESS patients) were enrolled to analyze. 5 participants in the control group were not included to analyze (3 cases failed a screening with CD4<200 cells/mm3 and 2 cases as diagnosis change).
Groups:
- Anti- TNF-a Treatment (SJS/TEN); Anti- TNF-a Treatment (DRESS): 1. Meet the conditions of inclusion and exclusion, seek the consent of the patient, and fill out the ICF
  2. Fill out the case report form
  3. Blood test and physiological assessment, and do TNF-alpha serum concentration and peripheral blood mononuclear spherical cDNA expression analysis
  4. Etanercept administration:
  The experimental group received the first dose of Etanercept (25 mg) i.v., followed by two doses per week and maintain 2 to 3 weeks
  anti-TNF a: 25mg BIW, SC
- Control Group (SJS/TEN); Control Group (DRESS): 1. Meet the conditions of inclusion and exclusion, seek the consent of the patient, and fill out the ICF
  2. Fill out the case report form
  3. Blood test and physiological assessment, and do TNF-alpha serum concentration and peripheral blood mononuclear spherical cDNA expression analysis
  4. Drug administration:
  The control group of drug delivery: systemic intravenous steroid therapy, the dose is equivalent to prednisolone 1-1.5 mg / kg / day, according to the treatment of 3-4 days gradually decreased dose.
Period: Overall Study
Arm/Group | Anti- TNF-a Treatment (SJS/TEN) | Control Group (SJS/TEN) | Anti- TNF-a Treatment (DRESS) | Control Group (DRESS)
Started | 48 | 43 | 22 | 22
Completed | 38 | 33 | 18 | 17
Not Completed | 10 | 10 | 4 | 5

BASELINE CHARACTERISTICS:
Population: A total of 135 SCAR patients (including 91 SJS/TEN cases and 44 DRESS cases) were enrolled to analyze.
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti- TNF-a Treatment (SJS/TEN) | Control Group (SJS/TEN) | Anti- TNF-a Treatment (DRESS) | Control Group (DRESS) | Total
Number analyzed (Participants) | 48 | 43 | 22 | 22 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 5 | 0 | 0 | 6
  Between 18 and 65 years | 35 | 15 | 17 | 11 | 78
  >=65 years | 12 | 23 | 5 | 11 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.73 (16.78) | 59.84 (24.20) | 53.95 (17.41) | 60.95 (20.39) | 56.53 (20.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 14 | 15 | 80
  Male | 20 | 20 | 8 | 7 | 55
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 48 | 43 | 22 | 22 | 135

OUTCOME MEASURES:

1. Primary Outcome: Skin Healing Time
Description: Healing was defined as complete re-epithelialization (i.e., the complete absence of erosions). We recorded the time taken by the skin to heal.
Time Frame: One to two months for SJS/TEN cases, and one to six months for DRESS cases.
Population: We determined if the enrolled participants had SJS/TEN and DRESS using the criteria and histopathological examinations.
Measure: Median (Full Range); unit: days
Arm/Group | Anti- TNF-a Treatment (SJS/TEN) | Control Group (SJS/TEN) | Anti- TNF-a Treatment (DRESS) | Control Group (DRESS)
Number analyzed (Participants) | 38 | 33 | 18 | 17
days | 13.75 [4 to 41] | 19 [7 to 42] | 40.5 [18 to 117] | 34 [9 to 165]
Statistical Analysis 1: Comparison: Anti- TNF-a Treatment (SJS/TEN) vs Control Group (SJS/TEN); For evaluating the time taken to heal skin erosion, the Kaplan-Meier product-limit estimates method was performed. Differences were considered statistically significant at P values of less than 0.05; Test type: Other; p = 0.01, Kaplan-Meier analysis — The p-value was analyzed for SJS/TEN participants with >10% body surface area detachment
Statistical Analysis 2: Comparison: Anti- TNF-a Treatment (DRESS) vs Control Group (DRESS); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.06, Kaplan-Meier analysis — This p-value was analyzed for DRESS participants

ADVERSE EVENTS:
Time Frame: one to two months
Description: The endpoints of serious adverse event and adverse event were assessed for three weeks after discharge.
Arm/Group | Anti- TNF-a Treatment (SJS/TEN) | Control Group (SJS/TEN) | Anti- TNF-a Treatment (DRESS) | Control Group (DRESS)
Serious Adverse Events (participants affected / at risk) | 5/48 | 9/43 | 2/22 | 5/22
Other Adverse Events (participants affected / at risk) | 15/48 | 19/43 | 8/22 | 8/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti- TNF-a Treatment (SJS/TEN) (N=48) | Control Group (SJS/TEN) (N=43) | Anti- TNF-a Treatment (DRESS) (N=22) | Control Group (DRESS) (N=22)
Sepsis (Infections and infestations) | 2 (2) | 4 (4) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper GI hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Stridor, vocal cord palsy (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti- TNF-a Treatment (SJS/TEN) (N=48) | Control Group (SJS/TEN) (N=43) | Anti- TNF-a Treatment (DRESS) (N=22) | Control Group (DRESS) (N=22)
Hypertension (Vascular disorders) | 6 (6) | 5 (5) | 3 (3) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (8) | 8 (8) | 4 (4) | 3 (3)
GI hemorrhage (grade 2) (Gastrointestinal disorders) | 1 (1) | 6 (6) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes